CLINICAL TRIAL: NCT04031742
Title: Phase 2b/3 Study to Assess the Efficacy and Safety of IBI306 in Subjects With Homozygous Familial Hypercholesterolemia.
Brief Title: A Study to Evaluate Safety and Efficacy of IBI306, a PCSK9 Monoclonal Antibody in Chinese Subjects With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI306A201
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12 [ Time Frame: Baseline and Week 12 ]
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: IBI306 (Experimental): Participants receive open-label IBI306 150 mg subcutaneously Q2W or 450 mg Q4W for 12 weeks.
  Interventions: Biological: IBI306
- Part 2: IBI306 (Experimental): Participants receive open-label 450 mg Q4W subcutaneously for 12 weeks.
  Interventions: Biological: IBI306

INTERVENTIONS:
Biological: IBI306 — Administered by subcutaneous injection
  Arms: Part 1: IBI306
Biological: IBI306 — Administered by subcutaneous injection
  Arms: Part 2: IBI306

SUMMARY:
A study to evaluate safety and efficacy of IBI306 in subjects with homozygous familial hypercholesterolemia.

DETAILED DESCRIPTION:
This is a phase 2b/3 study to assess the efficacy and safety of IBI306 in subjects with homozygous familial hypercholesterolemia. Part 1 is an open-label, two-arm, multicenter pilot study to evaluate efficacy and safety of IBI306 in subjects with homozygous familial hypercholesterolemia. Part 2 is an open-label, single-arm, multicenter study to evaluate efficacy and safety of IBI306 in subjects with homozygous familial hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 to ≤ 80 years of age
2. Diagnosis of homozygous familial hypercholesterolemia
3. LDL cholesterol ≥ 130 mg/dL (3.4mmol/L)
4. Triglyceride ≤ 400 mg/dL (4.5 mmol/L)
5. Bodyweight of ≥ 40 kg at screening

Exclusion Criteria:

1. History of liver transplant
2. Uncontrolled hypertension
3. Moderate to severe renal dysfunction
4. Active liver disease or hepatic dysfunction
5. Known sensitivity to any of the products to be administered during dosing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Part 1: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C). | Baseline and Week 12
Part 2: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) | Baseline and Week 12

OTHER OUTCOMES:
Number of investigational product-related adverse events. | Baseline and Week 12
Number of ADA and Nab. | Baseline and Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China